CLINICAL TRIAL: NCT04604314
Title: Clinical Performance of Alternative Preparation Designs for Chairside CAD/CAM Fabricated Advanced Lithium Disilicate EndoCrowns
Brief Title: Alternative EndoCrowns Designs for Chairside CAD/CAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Principal Investigator, Dennis J. Fasbinder, DDS, Clinical Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00172803
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Endodontically Treated Teeth
Keywords: Ceramic; Crown; Endocrown
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Endocrown Onlay Restoration (Experimental): Endocrown onlay preparation = Buccal and lingual walls are intact with an occlusal-gingival height at least equal to half the original crown height of the tooth. Remaining buccal and lingual walls maintain a thickness ≥ 2.0 mm.
  Interventions: Device: CEREC Tessera
- Endocrown Shoulder Restorations (Experimental): Endocrown shoulder preparation = Buccal and/or lingual walls are less than half the original occlusal-gingival height of the tooth or the buccal or lingual surfaces were previously prepared axially due to a prior restoration.
  Interventions: Device: CEREC Tessera

INTERVENTIONS:
Device: CEREC Tessera — Full ceramic endocrown restorations will be made from the high strength ceramic, CEREC Tessera

SUMMARY:
This investigation will be a longitudinal clinical trial to study the association of preparation design on the internal and marginal adaptation of the resulting restorations and the long-term clinical performance of chairside CAD/CAM endocrown restorations. Advanced lithium disilicate chairside CAD/CAM endocrowns (CEREC Tessera/Dentsply Sirona) will be adhesively bonded using a selective enamel etch technique with a universal adhesive (Prime and Bond Elect/Dentsply Sirona) and a dual cure resin adhesive cement (Calibra Ceram/Dentsply Sirona). All restorations will be followed over five years of clinical service.

DETAILED DESCRIPTION:
Endodontically treated teeth commonly present with extensive tooth structure loss due to caries, trauma, prior restorative treatment, and the endodontic access. These structural deficiencies lead to an increase in cusp deflection, crown fractures, microleakage, and decreased sensory feedback during function which greatly increases the possibility of tooth fracture.As a result, endodontically treated teeth require a full cuspal coverage restoration to prevent microleakage, restore function, and provide cuspal protection against tooth fracture. The most common restoration for endodontically treated teeth is core build-up, with or without a post, and full coverage crown.

This process requires multiple appointments with many technical steps ultimately leading to more chair time, treatment cost, and potential iatrogenic damage to the tooth. An alternative treatment is the endocrown, which utilizes the internal walls of the pulp chamber for macroretention and incorporates the core and crown in a monolithic restoration. The restoration is fabricated utilizing chairside CAD/CAM technology and is adhesively bonded to the tooth with resin cement. The EndoCrown restoration is more conservative relative to tooth structure loss, less expensive, and requires less chair time to complete when compared to conventional treatment while having comparable clinical longevity in molar teeth.

This investigation will be a longitudinal clinical trial to study the association of preparation design on the internal and marginal adaptation of the resulting restorations and the long-term clinical performance of chairside CAD/CAM endocrown restorations. Advanced lithium disilicate chairside CAD/CAM endocrowns (CEREC Tessera/Dentsply Sirona) will be adhesively bonded using a selective enamel etch technique with a universal adhesive (Prime and Bond Elect/Dentsply Sirona) and a dual cure resin adhesive cement (Calibra Ceram/Dentsply Sirona). All restorations will be followed over five years of clinical service.

ELIGIBILITY:
Inclusion Criteria:

1. Subject in need of final restoration following molar endodontic therapy
2. Subject age 18 or above -

Exclusion Criteria:

1. Teeth with remaining symptoms following endodontic therapy
2. Teeth which have experienced endodontic complications to include treated perforations, internal or external resorption, or separated endodontic files.
3. Teeth with exposure of the root canal filling material to the oral environment for greater than two weeks
4. Teeth diagnosed with symptoms of incomplete tooth fracture
5. Teeth with no adjacent or opposing tooth
6. Teeth serving as an abutment for fixed or removable dental prostheses
7. Subjects with uncontrolled bruxism or parafunctional habits
8. Subject has known allergies to any product used in this study
9. Subject will not be available for the study duration of 5 years
10. Subjects with significant untreated dental disease to include periodontitis and rampant caries
11. Women who self-report that they are pregnant or lactating

    -

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Restoration failure | from delivery of the crown up to 5 years
  Restoration failure is scored by visual loss of the crown from the tooth requiring replacement of the study crown with a new crown at any time between delivery and five years.

SECONDARY OUTCOMES:
Restoration loss of retention | from delivery of crown up to 5 years
  Loss of retention is measured as visual detachment or dislodgment of the crown from the tooth without fracture of the crown requiring recementation of the crown.
Margin staining | from delivery of crown up to 5 years
  Margin staining is categorized based on modified US Public Health Service criteria using a four point scale where 1 is no staining and 4 is penetrating stain involving more than 50% of the margin.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Fasbinder, DDS, Principal Investigator — University of Michigan
Locations (1):
- School os Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No